CLINICAL TRIAL: NCT00948298
Title: The Effect of Cholecalciferol (Vitamin D3) on Vascular Function and Cardiovascular Risk Factors
Brief Title: Effect of Vitamin D3 on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, David Martins, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB#08-05-2170-01; U54RR022762 (NIH)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Vitamin D Deficiency
Keywords: cardiovascular disease; vitamin D; african american; low vitamin D levels
MeSH Terms: conditions — Vitamin D Deficiency; Cardiovascular Diseases | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vitamin D (Experimental)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Two 50,000 IU tablets of oral Vitamin D3 will be given every 4 weeks.
  Arms: Vitamin D
Drug: Placebo — Two tablets of oral placebo (microcrystalline cellulose),matching in appearance to the Vitamin D3, will be given every 4 weeks.
  Arms: Placebo

SUMMARY:
Vitamin D is a natural nutrient. A little comes from our normal daily diet. Most of it comes from our skin after we have been in sunlight. If we have darker skin, we make less vitamin D. Vitamin D balances the calcium in our body. If our vitamin D levels get too low, it can cause health problems. It may increase our chance of getting high blood pressure or diabetes. Another problem we may have if our vitamin D levels are low is that our blood vessels may not work normally. These are important health problems for anyone. Because African Americans have darker skin, they are more likely than most other racial/ethnic groups to have low vitamin D levels. This study will look at treating African Americans with low vitamin D levels.

The goal of this study is to see how vitamin D helps blood vessels work. The investigators will do this study in African Americans who are overweight, have high blood pressure and have low vitamin D levels. The investigators will see if getting the vitamin D level to a normal value will improve how blood vessels work. The dose of vitamin D that will be given in this study is a high dose that is given to people with low vitamin D levels.

DETAILED DESCRIPTION:
Cardiovascular Disease (CVD) and related disorders remain the leading cause of death in the nation. Hypovitaminosis D has been linked not only to several cardiovascular (CV) risk factors including hypertension, diabetes, obesity but also to increased rates of CVD. Thus,hypovitaminosis D presents a common pathway for a select subgroup with a clustering of CV risk factors in a profile that is predominant among ethnic minorities. Indeed, hypovitaminosis D is highly prevalent with an estimated 55% of the US adult population having levels at or below 30 ng/ml, and over 80% of African Americans having suboptimal values. Thus, we propose a twelve week randomized double-blind, placebo controlled pilot trial to assess the effect on vascular function and CV risk factors of 100,000 IU Vitamin D3 given every 4 weeks to overweight, hypertensive African-Americans with hypovitaminosis D. To our knowledge, the proposed project is the first to assess the effect of 'high-dose' Vitamin D3 administration on vascular function.We believe this study is also the first to examine the impact at a molecular level of Vitamin D3 repletion on the key mediators of cardio-metabolic pathways in humans. If our study results support our working hypothesis, we will be positioned to propose a larger scale study to detect a therapeutic effect on more definitive, clinical cardiovascular endpoints across a more diverse population.

Objectives:

1. Assess the role of Vitamin D3 treatment on vascular function in high risk subjects.

Primary Outcome: The primary outcome variable is pulse wave velocity (PWV, unit - m/s) for vascular stiffness assessed by radial artery tonometry (via SphygmoCor). The hypothesis for the primary analysis is that a greater increase in the PWV will occur in the Vitamin D3 treatment group than in the placebo group.

Secondary Outcome: Vascular/endothelial function as determined by measuring non-invasive vascular finger plethysmography (via EndoPat). Additional surrogates to be assessed as secondary markers of vascular/endothelial function include sitting and 24 hour ambulatory blood pressure measurements and spot urine protein/creatinine ratio.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18-70 years of age and self-identified as African-American or Black
* Hypertension
* If a potential study patient is not on treatment, their systolic blood pressure (SBP) must be > 130 mmHg, or diastolic blood pressure (DBP) > 85 mmHg, and SBP must be <160 mmHg and DBP must be < 105 mmHg.
* If a potential study patient is on treatment then the SBP must be <160 mmHg and DBP must be < 105 mmHg
* Screening Vitamin D (D2 and D3 level) between 10 and 25 ng/ml (normal level > 30 ng/ml)
* Body mass index (BMI) > 25 kg/m2

Exclusion Criteria:

* Poorly controlled high blood pressure (SBP >160 mmHg or DBP > 105 mmHg)
* Diabetes (fasting blood sugar > 125 mg/dl, or HbA1c > 6.5%)
* Screening Vitamin D (D2 and D3 level) < 10 ng/ml or > 25 ng/ml
* Estimated glomerular filtration rate (eGFR) < 45 ml/min
* Evidence of disease resulting in hypercalcemia
* History of kidney stones
* History of drug, alcohol, or illicit substance abuse within the past 6 months
* History of another chronic disease which the investigator feels should preclude the subject from entering the study
* Liver function tests (LFTs) greater than twice the upper limit of normal
* Subjects requiring chronic use of nonsteroidal anti-inflammatory drugs, aspirin, or other drugs that may affect the measurement of reactive oxidative species
* Subjects requiring treatment with other vitamin D preparations containing more than 400 IU of vitamin D
* Subjects requiring chronic use of immunosuppressive therapy or corticosteroids
* Recent (< 6 months) myocardial infarction, stroke, or hospitalization for congestive heart failure
* Allergy/intolerance: known allergy to oral vitamin D or microcrystalline cellulose

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Martins, MD, Principal Investigator — Charles Drew University of Medicine and Science

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Two tablets of oral placebo (microcrystalline cellulose),matching in appearance to the Vitamin D3 will be given every 4 weeks.
- Vitamin D: Two 50,000 IU tablets of oral Vitamin D3 given every 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 65 | 65
Completed | 55 | 60
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Customized [Count of Participants; unit: Participants]
  18-39 years | 10 | 10 | 20
  40-59 years | 47 | 45 | 92
  60 years and above | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 38 | 41 | 79
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 65 | 130
Body Mass Index, Categorical [Count of Participants; unit: Participants]
  25.0-29.9 kg/m^2 | 18 | 12 | 30
  >30 kg/m^2 | 47 | 53 | 100
Waist Circumference Groups [Count of Participants; unit: Participants]
  Low (<102 cm for male and <88 cm for female) | 17 | 12 | 29
  High (>=102 cm for male and >=88 cm for female) | 48 | 53 | 101
Blood Pressure (Systolic) [Mean (Standard Deviation); unit: mmHg] | 128.5 (15.2) | 125.2 (16.1) | 126.8 (15.7)
Blood Pressure (Diastolic) [Mean (Standard Deviation); unit: mmHg] | 84.5 (10.5) | 80.9 (11.4) | 82.7 (11.1)
Augmentation Index [Mean (Standard Deviation); unit: percentage of central pulse pressure] — Augmentation Index (Aix) is the percentage of central pulse pressure (central systolic minus diastolic pressure) attributable to the reflection of the pulse wave at arterial bifurcation points and interface of the large arteries and small resistance arteries. It is the index of aortic pressure wave reflection, defined as the ratio of augmented ascending aortic pressure (generated backward traveling pressure waves) to the central pulse pressure at the aortic root: where (Ps - Pi) / (Ps - Pd) Ps = peak systolic pressure, Pi = pressure at reflection point, and Pd = minimum diastolic pressure.
  percentage of central pulse pressure | 31.0 (12.0) | 28.2 (11.2) | 29.6 (11.6)
Urine Isoprostane [Mean (Standard Deviation); unit: ng/mg] | 14.9 (15.8) | 14.4 (11.6) | 14.6 (13.8)
Serum 25(OH)D Level [Mean (Standard Deviation); unit: nmol/L] | 16.5 (5.0) | 17.0 (5.2) | 16.8 (5.1)
Serum Calcium Level [Mean (Standard Deviation); unit: mg/dl] | 9.3 (0.4) | 9.4 (0.3) | 9.4 (0.4)
Intact Parathyroid Hormone (PTH) Level [Mean (Standard Deviation); unit: pmol/L] | 49.9 (33.6) | 43.4 (19.9) | 46.7 (27.7)

OUTCOME MEASURES:

1. Primary Outcome: Pulse Wave Velocity for Vascular Stiffness
Description: The primary outcome variable is pulse wave velocity (PWV) for vascular stiffness. The hypothesis is that a greater decrease in the PWV will occur with the Vitamin D3 treatment. PWV is the speed at which the arterial pulse wave travels through the arteries in the cardiovascular system. It is considered the gold standard for the assessment of arterial elastance (stiffness) and determined by radial artery applanation tonometry using the SphygmoCor device.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 65 | 65
m/s | 29.3 (11.0) | 27.6 (11.0)

2. Secondary Outcome: Changes in Sitting and 24 Ambulatory Blood Pressure
Description: Improved vascular function as determined by measuring sitting and 24 Hour Ambulatory Blood Pressure.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 65 | 65
mmHg
  Blood Pressure (Systolic) | 125.8 (13.3) | 126.9 (15.0)
  Blood Pressure (Diastolic) | 82.2 (9.2) | 81.1 (12.0)
  24 Hour Blood Pressure (Systolic) | 128.4 (14.0) | 127.4 (16.4)
  24 Hour Blood Pressure (Diastolic) | 83.9 (10.1) | 82.0 (11.6)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Groups:
- Placebo: Two tablets of oral placebo (microcrystalline cellulose), matching in appearance to the Vitamin D3, will be given every 4 weeks.
Arm/Group | Placebo | Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 4/65 | 4/65
Other Adverse Events (participants affected / at risk) | 12/65 | 14/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Vitamin D (N=65)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Post Biopsy Bleeding at Wound Site (Surgical and medical procedures) | 1 (2) | 0 (0)
Pituitary Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Elevated Blood Pressure (Vascular disorders) | 1 (3) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (4) | 0 (0)
Atypical Chest Pain (Cardiac disorders) | 0 (0) | 1 (3)
Syncope (General disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Vitamin D (N=65)
Hemoglobin = 9.6 G/DL (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
High Platelet Count = 493 Thousand/UL (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hematocrit = 30.2% (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated WBC = 14.9 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Low White Blood Cell Count = 2.9 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral Edema, Left and Right Feet (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low Platelet Count = 107 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated Platelet = 456 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Elevated iPTH = 213 (Endocrine disorders) | 1 (1) | 0 (0)
Elevated iPTH = 236 (Endocrine disorders) | 1 (1) | 0 (0)
Elevated SGOT = 103 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated SGPT = 106 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gallbladder Removed (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infection at Biopsy Site (Infections and infestations) | 1 (1) | 0 (0)
Phosphate = 5.0 MG/DL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
iPTH = 7 PG/ML (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Back Discomfort from Car Accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Hip Pain; Osteoarthritis Flare Up; Exacerbation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pituitary Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Creatinine = 1.44 MG/DL (Renal and urinary disorders) | 1 (1) | 0 (0)
Creatinine Random Urine = 461.3 (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin Sensitivity to Adhesive Tape Post Biopsy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elevated Blood Pressure (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No